CLINICAL TRIAL: NCT05204342
Title: Evaluation of Prognostic Factors for Tubo-ovarian Cancer in France: Surgical Thresholds, Geographical Distance, Age and Therapeutic Sequence
Brief Title: Evaluation of Prognostic Factors for Tubo-ovarian Cancer in France
Acronym: Pro-TOCa
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0742
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian or Tubal Cancer; Upfront surgery; surgical thresholds
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the following prognostic factors in France, based on national quotation data: volume per center, patient age, geographic distance from a clinical center, delay for chemotherapy,Upfront surgery.

ELIGIBILITY:
Inclusion criteria:

* - Diagnosic of Ovarian or Tubal Cancer C56 et C570
* +/-
* Carcinose péritonéale C786
* Tumueur maligne secondaire de la plèvre C782,
* Tumueur maligne secondaire des ganglions C770 à C779,
* Tumueur maligne secondaire du foie C787,
* Tumueur maligne secondaire du péritoine C786

Exclusion criteria:

* autres causes de :
* Carcinose péritonéale C786
* Tumueur maligne secondaire de la plèvre C782,
* Tumueur maligne secondaire des ganglions C770 à C779,
* Tumueur maligne secondaire du foie C787,
* Tumueur maligne secondaire du péritoine C786

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women treated for tubo-ovarian cancer in France between 2012 and 2016
Sampling Method: Non-Probability Sample
Enrollment: 22500 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
To study the prognostic effect of the volume of activity | at 5 years
  To study the prognostic effect of the volume of activity per center on the risk of recurrence
Verify that the therapeutic sequence | at 5 years
  Verify that the therapeutic sequence of primary surgery and secondary chemotherapy is a good prognostic factor for overall and specific survival at 5 years

SECONDARY OUTCOMES:
Verify that delay in initiation of chemotherapy beyond 4 weeks | at 5 years
  Verify that delay in initiation of chemotherapy beyond 4 weeks after surgery is a poor prognostic element on overall and specific survival at 5 years
Verify that age is a poor prognostic element | at 5 years
  Verify that age is a poor prognostic element for overall and specific survival at 5 years
Verify that geographic distance | at 5 years
  Verify that geographic distance from a clinical center is a poor prognostic element for overall and specific survival at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Martha DURAES, Md, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC